CLINICAL TRIAL: NCT00062244
Title: Phase I/II Study of G3139 (Genasense) in Patients With Waldenstrom's Macroglobulinemia
Brief Title: Oblimersen in Treating Patients With Relapsed or Refractory Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01437; MC0285; MAYO-MC0285; NCI-5826; CDR0000304634; N01CM17104 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — oblimersen

ARMS (1):
- Arm I (Experimental): Phase I: Patients receive oblimersen IV continuously on days 1-7. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 1-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Phase II: Patients receive treatment as in phase I at the MTD of oblimersen. Patients are followed every 3 months for 2 years.
  Interventions: Biological: oblimersen sodium

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense

SUMMARY:
This phase I/II trial is studying the side effects and best dose of oblimersen and to see how well it works in treating patients with relapsed or refractory Waldenstrom's macroglobulinemia. Biological therapies such as oblimersen may interfere with the growth of the cancer cells and slow or stop the growth of Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) and recommended dosing for Genasense in patients with relapsed or refractory WM following prior chemotherapy. (Phase I) II. To determine the response rate to Genasense in patients with relapsed or refractory WM following prior chemotherapy.

III. To determine the safety of Genasense in patients with relapsed or refractory WM following prior chemotherapy.

IV. To describe possible clinical benefit from Genasense treatment of relapsed or refractory WM including duration of response, survival, erythropoietin use, improvement in hemoglobin > 11 g/dl, and Improvement in platelet count > 100,000/mm^3.

OUTLINE: This is a multicenter, dose-escalation study.

Phase I: Patients receive oblimersen IV continuously on days 1-7. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 1-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive treatment as in phase I at the MTD of oblimersen. Patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Waldenstrom's macroglobulinemia (WM) confirmed by both of the following:

  * Bone marrow lymphoplasmacytosis with greater than 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy
  * Measurable disease, defined by quantitative IgM monoclonal protein greater than 1,000 mg/dL
* Symptomatic relapsed or refractory disease requiring therapy, defined by at least 1 of the following:

  * Impaired bone marrow function due to disease infiltration as demonstrated by any of the following:

    * Hemoglobin less than 11 g/dL
    * Requires epoetin alfa therapy to maintain hemoglobin of at least 11 g/dL
    * Platelet count less than 100,000/mm^3
  * Symptomatic bulky lymphadenopathy
  * Symptoms attributable to hyperviscosity (e.g., nose bleeding, gingival bleeding, or retinal hemorrhage) or serum viscosity level relative to water greater than 4
* Received at least 1 prior chemotherapy regimen which included chlorambucil, cyclophosphamide, fludarabine, cladribine, or pentostatin
* No secondary leukemia or history of antecedent hematologic disorder (e.g., myelodysplasia) prior to initial onset of WM
* Performance status - ECOG 0-2
* Not specified
* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 50,000/mm^3*
* No bleeding disorder
* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST less than 1.5 times ULN
* Albumin at least 2.5 g/dL
* PT no greater than 1.5 times ULN
* INR no greater than 1.3
* PTT no greater than 1.5 times ULN
* No history of chronic hepatitis or cirrhosis
* Creatinine no greater than 2 times ULN
* No uncontrolled congestive heart failure
* No active symptoms of coronary artery disease, including the following:

  * Uncontrolled arrhythmias
  * Recurrent chest pain despite prophylactic medication
* No New York Heart Association class III or IV heart disease
* No grade 2 or greater cardiovascular signs and symptoms within the past 4 weeks
* HIV negative
* Direct Coombs' test negative
* No autoimmune thrombocytopenia
* No uncontrolled serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate venous access for 7-day continuous infusion of study drug
* Intellectual, emotional, and physical ability to maintain an ambulatory infusion pump
* No other cancer except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other cancer from which the patient has been disease-free for at least 5 years
* No known hypersensitivity to phosphorothioate-containing oligonucleotides
* No uncontrolled seizure disorder
* More than 21 days since prior immunotherapy for WM
* More than 21 days since prior cytokine, biologic, or vaccine therapy for WM
* More than 8 weeks since prior plasmapheresis or plasma exchange
* No prior allogeneic stem cell transplantation
* No concurrent plasmapheresis or plasma exchange
* See Disease Characteristics
* No concurrent corticosteroid therapy
* More than 21 days since prior radiotherapy for WM
* More than 21 days since prior major surgery for WM
* No prior organ allograft
* Recovered from all prior therapy
* More than 21 days since other prior therapy for WM
* No other concurrent investigational therapy
* No concurrent immunosuppressive drugs
* No concurrent therapeutic anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-05; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by the number of dose-limiting toxicity incidents graded according to CTC standard toxicity (Phase I) | 21 days
  Hematologic dose-limiting toxicity measures will be assessed using the continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization.

SECONDARY OUTCOMES:
Adverse events that are classified as either possibly, probably, or definitely related to study treatment (Phase II) | Up to 2 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Proportion of overall confirmed responses (CR + PR) associated with G3139 (Phase II) | 6 months
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time to progression | Time from registration to the time of progression, assessed up to 2 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Overall survival | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Duration of response | From the documentation of response until the date of progression, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Morie Gertz, Principal Investigator — Mayo Clinic
Locations (8):
- United States (8):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Howard University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin